CLINICAL TRIAL: NCT04137380
Title: A Single-Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of LY3074828 in Healthy Chinese Subjects
Brief Title: A Study of Mirikizumab in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 16766; I6T-MC-AMBD (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Results first posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2023-05

CONDITIONS: Healthy
MeSH Terms: interventions — mirikizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Mirikizumab - Intravenous (IV) (Experimental): Participants received a single dose of 300 milligram (mg), 600 mg and 1200 mg mirikizumab administered IV using a forearm vein infused over at least 30 minutes, 60 minutes and 2 hours.
  Interventions: Drug: Mirikizumab - IV
- Placebo - IV (Placebo Comparator): Participants received a single dose of placebo administered IV using a forearm vein.
  Interventions: Drug: Placebo - IV
- Mirikizumab - Subcutaneous (SC) (Experimental): Participants received a single dose of 200 mg, 400 mg mirikizumab administered SC as 2 injections, 1 into the skinfold of each lower abdominal wall quadrant (left and right).
  Interventions: Drug: Mirikizumab - SC
- Placebo - SC (Placebo Comparator): Participants received a single dose of placebo administered SC as 2 injections, 1 into the skinfold of each lower abdominal wall quadrant (left and right).
  Interventions: Drug: Placebo - SC

INTERVENTIONS:
Drug: Mirikizumab - IV — Administered IV
  Other Names: LY3074828
  Arms: Mirikizumab - Intravenous (IV)
Drug: Mirikizumab - SC — Administered SC
  Other Names: LY3074828
  Arms: Mirikizumab - Subcutaneous (SC)
Drug: Placebo - IV — Administered IV
  Arms: Placebo - IV
Drug: Placebo - SC — Administered SC
  Arms: Placebo - SC

SUMMARY:
The main purpose of this study is to evaluate the safety of the study drug known as mirikizumab. The study will investigate how the body processes the study drug. It will last up to about 4 months for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Native Chinese (all 4 biological grandparents and both biological parents to be Chinese origin)
* Have a body mass index (BMI) of 18.0 to 32.0 kilograms per square meter (kg/m²), inclusive, at time of screening
* Have clinical laboratory test results within normal reference range for the investigative site or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Have venous access sufficient to allow for blood sampling and administration of investigational product (IP) or placebo
* Are reliable and willing to be available for the duration of the study and are willing to follow study procedures
* Are able and willing to give signed informed consent

Exclusion Criteria:

* Are currently enrolled in a clinical study involving an IP or any other type of medical research judged not to be scientifically or medically compatible with this study
* Have participated in a clinical trial involving an IP within 30 days or 5 half-lives (whichever is longer) prior to screening. If the clinical trial involved treatment with biologic agents (such as monoclonal antibodies, including marketed drugs), at least 3 months or 5 half-lives (whichever is longer) should have elapsed prior to Day 1
* Have known allergies to LY3074828, humanized monoclonal antibodies, related compounds or any components of the formulation, or history of significant atopy
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen or positive hepatitis B core antibody
* Have had symptomatic herpes zoster within 3 months of screening
* Show evidence of active or latent tuberculosis (TB), as documented by medical history, examination, chest X-rays (posterior/anterior and lateral), and TB testing (positive or indeterminate for QuantiFERON® -TB Gold test or T-Spot. 1 retest permitted following indeterminate result); or have had household contact with a person with active TB, unless appropriate and documented prophylaxis treatment has been given. Participants with any history of active TB are excluded from the study, regardless of previous or current TB treatments.
* Have received live vaccine(s), including attenuated live vaccines and those administered intranasally, within 8 weeks of screening, or intend to during the study
* Are immunocompromised
* Have clinically significant multiple or severe drug allergies, or intolerance to topical corticosteroids, or severe post treatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear immunoglobulin A dermatosis, toxic epidermal necrolysis, or exfoliative dermatitis)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2020-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- China (2):
  - Shanghai Xuhui Central Hospital, Xuhui District, Shanghai Municipality
  - Peking University First Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Intravenous (IV): Participants received a single dose of placebo administered IV using a forearm vein.
- 300 Milligram (mg) Mirikizumab IV: Participants received a single dose of 300 mg mirikizumab administered IV using a forearm vein infused over at least 30 minutes.
- 600 mg Mirikizumab IV: Participants received a single dose of 600 mg mirikizumab administered IV using a forearm vein infused over at least 60 minutes.
- 1200 mg Mirikizumab IV: Participants received a single dose of 1200 mg mirikizumab administered IV using a forearm vein infused over at least 2 hours.
- Placebo Subcutaneous (SC): Participants received a single dose of placebo administered SC as 2 injections, 1 into the skinfold of each lower abdominal wall quadrant (left and right).
- 200 mg Mirikizumab SC: Participants received a single dose of 200 mg mirikizumab administered SC as 2 injections, 1 into the skinfold of each lower abdominal wall quadrant (left and right).
- 400 mg Mirikizumab SC: Participants received a single dose of 400 mg mirikizumab administered SC as 4 injections, 1 into the skinfold of each lower abdominal wall quadrant (left and right).
Period: Overall Study
Arm/Group | Placebo Intravenous (IV) | 300 Milligram (mg) Mirikizumab IV | 600 mg Mirikizumab IV | 1200 mg Mirikizumab IV | Placebo Subcutaneous (SC) | 200 mg Mirikizumab SC | 400 mg Mirikizumab SC
Started | 6 | 10 | 10 | 10 | 4 | 10 | 10
Received at Least One Dose of Study Drug | 6 | 10 | 10 | 10 | 4 | 10 | 10
Completed | 6 | 10 | 10 | 9 | 4 | 10 | 10
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Placebo IV: Participants received a single dose of placebo administered IV using a forearm vein.
- 300 mg Mirikizumab IV: Participants received a single dose of 300 mg mirikizumab administered IV using a forearm vein infused over at least 30 minutes.
- Placebo SC: Participants received a single dose of placebo administered SC as 2 injections, 1 into the skinfold of each lower abdominal wall quadrant (left and right).
- Total: Total of all reporting groups
Arm/Group | Placebo IV | 300 mg Mirikizumab IV | 600 mg Mirikizumab IV | 1200 mg Mirikizumab IV | Placebo SC | 200 mg Mirikizumab SC | 400 mg Mirikizumab SC | Total
Number analyzed (Participants) | 6 | 10 | 10 | 10 | 4 | 10 | 10 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.0 (6.2) | 32.4 (6.4) | 31.7 (5.3) | 36.5 (6.1) | 25.0 (5.0) | 33.9 (7.2) | 31.8 (6.2) | 32.0 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 4 | 4 | 0 | 5 | 4 | 23
  Male | 4 | 6 | 6 | 6 | 4 | 5 | 6 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 10 | 10 | 10 | 4 | 10 | 10 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 10 | 10 | 10 | 4 | 10 | 10 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 6 | 10 | 10 | 10 | 4 | 10 | 10 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Drug-Related Treatment-Emergent Adverse Events (TEAEs)
Description: Drug-related TEAEs are any untoward medical occurrence that either occurs or worsens at any time after treatment baseline, and in the opinion of the investigators is possibly related to study drug. A summary of serious adverse events (SAEs) and other non-serious adverse events (NSAEs), regardless of whether or not they were possibly related to study drug, is located in the Reported Adverse Event section.
Time Frame: Baseline through Day 85
Population: All randomized participants who received at least one dose of study drug and have at least one postdose safety assessment.
Measure: Number; unit: participants
Arm/Group | Placebo IV | 300 mg Mirikizumab IV | 600 mg Mirikizumab IV | 1200 mg Mirikizumab IV | Placebo SC | 200 mg Mirikizumab SC | 400 mg Mirikizumab SC
Number analyzed (Participants) | 6 | 10 | 10 | 10 | 4 | 10 | 10
participants | 1 | 3 | 4 | 1 | 1 | 0 | 0

2. Primary Outcome: Visual Analog Scale (VAS) Pain Score for Subcutaneous Injection Site
Description: The injection pain VAS score is a participant administered single item scale designed to measure pain using a 0-100 millimeter (mm) horizontal VAS. The severity of pain was categorized by VAS pain score as: no pain (0), mild pain ≤ 30, moderate pain (>30 and ≤70), and severe pain (>70). Overall severity of participant's pain is indicated by placing a single mark on the horizontal 100 mm scale from 0 mm (no pain) to 100 mm (worst imaginable pain).
Time Frame: 0 min, 0.25 hours (h), 0.5 h, 1 h, 2 h and 4 h post first injection
Population: All randomized participants who received at least one dose of study drug and have at least one postdose safety assessment. As per statistical analysis plan, VAS pain score was analyzed only for SC dose.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Placebo SC | 200 mg Mirikizumab SC | 400 mg Mirikizumab SC
Number analyzed (Participants) | 4 | 10 | 10
millimeter (mm)
  0 min | 36.5 (36.3) | 30.8 (29.5) | 42.4 (26.0)
  0.25 h | 3.5 (3.3) | 2.9 (3.7) | 10.6 (20.2)
  0.5 h | 2.3 (2.6) | 1.9 (3.4) | 9.5 (23.1)
  1 h | 1.0 (0.8) | 1.6 (1.9) | 2.0 (1.8)
  2 h | 1.8 (1.0) | 1.2 (1.5) | 2.0 (2.0)
  4 h | 1.0 (0.8) | 1.0 (1.2) | 2.1 (2.6)

3. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Mirikizumab
Description: PK: Cmax of Mirikizumab was evaluated.
Time Frame: Pre-dose, [end of infusion (EOI) IV only], Day 1: 6 hours (h), Day 2, Day 4, Day 8, Day 11 (SC only), Day 15, Day 22, Day 29, Day 43, Day 57, Day 71, and Day 85 postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (μg/mL)
Arm/Group | 300 mg Mirikizumab IV | 600 mg Mirikizumab IV | 1200 mg Mirikizumab IV | 200 mg Mirikizumab SC | 400 mg Mirikizumab SC
Number analyzed (Participants) | 9 | 10 | 9 | 10 | 10
microgram per milliliter (μg/mL) | 145 (7) | 266 (16) | 511 (10) | 14.9 (28) | 23.1 (44)

4. Secondary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-∞]) of Mirikizumab
Description: PK: AUC(0-∞) of Mirikizumab was evaluated.
Time Frame: as for outcome 3
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*day per milliliter (μg*day/mL)
Arm/Group | 300 mg Mirikizumab IV | 600 mg Mirikizumab IV | 1200 mg Mirikizumab IV | 200 mg Mirikizumab SC | 400 mg Mirikizumab SC
Number analyzed (Participants) | 9 | 10 | 9 | 10 | 10
microgram*day per milliliter (μg*day/mL) | 936 (12) | 2030 (12) | 3320 (23) | 263 (29) | 421 (46)

5. Secondary Outcome: PK: AUC From Time Zero to Time T, Where T is the Last Sample With a Measurable Concentration (AUC[0-tlast]) of Mirikizumab
Description: PK: AUC(0-tlast) of Mirikizumab was evaluated.
Time Frame: as for outcome 3
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*day/mL
Arm/Group | 300 mg Mirikizumab IV | 600 mg Mirikizumab IV | 1200 mg Mirikizumab IV | 200 mg Mirikizumab SC | 400 mg Mirikizumab SC
Number analyzed (Participants) | 5 | 10 | 8 | 7 | 10
μg*day/mL | 964 (15) | 2010 (12) | 3300 (24) | 248 (34) | 417 (46)

ADVERSE EVENTS:
Time Frame: Up To 85 Days
Description: All randomized participants who received at least one dose of study drug and have at least one postdose safety assessment.
Arm/Group | Placebo IV | 300 mg Mirikizumab IV | 600 mg Mirikizumab IV | 1200 mg Mirikizumab IV | Placebo SC | 200 mg Mirikizumab SC | 400 mg Mirikizumab SC
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/10 | 0/10 | 0/10 | 0/4 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/10 | 0/10 | 0/10 | 0/4 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 5/6 | 7/10 | 9/10 | 3/10 | 3/4 | 4/10 | 5/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo IV (N=6) | 300 mg Mirikizumab IV (N=10) | 600 mg Mirikizumab IV (N=10) | 1200 mg Mirikizumab IV (N=10) | Placebo SC (N=4) | 200 mg Mirikizumab SC (N=10) | 400 mg Mirikizumab SC (N=10)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Animal scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood uric acid increased (Investigations) | 1 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Menstruation delayed (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis hypertrophic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 120 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2020-06-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT04137380/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/80/NCT04137380/SAP_001.pdf